CLINICAL TRIAL: NCT04391829
Title: Detection of SARS-CoV-2 in Semen of COVID-19 Positive Males
Acronym: COVIDSPERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVIDSPERM
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Sars-CoV2; Corona Virus Infection; Semen
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-CoV-2 positive men (Experimental): Men who are tested positive for SARS-CoV-2 by PCR testing on nasopharyngeal swab.
  Interventions: Diagnostic Test: Ejaculated semen sample

INTERVENTIONS:
Diagnostic Test: Ejaculated semen sample — SARS-CoV-2 positive men will be asked to give an ejaculated semen sample, within the seven days after positive testing. Semen samples will be performed every 7 days, until 2 semen PCR tests are negative and will be retested after 3 months.

SUMMARY:
The objectives of the study, are to describe detection of SARS-CoV-2 in the semen of COVID-19 positive patients, the duration of positive semen and to investigate the impact on semen quality, thereby providing insights into the early impact on male reproductive function.

DETAILED DESCRIPTION:
SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), a novel coronavirus reported in late December 2019 in Wuhan, China, has spread world-wide with over 1,000,000 coronavirus disease 2019 (COVID-19) cases reported. New developments in molecular virology and immunobiology of SARS-CoV-2, improve our understanding about COVID-19 prevention, management, and possible long-term effects. Although viral transmission occurs predominantly through respiratory droplets, SARS-CoV-2 has been isolated in blood samples and feces from COVID-19 patients, raising questions about viral shedding in other bodily fluids, including semen, as well as alternative modes of transmission.

The objectives are to describe detection of SARS-CoV-2 in the semen of COVID-19 positive patients, the duration of positive semen and to investigate the impact on semen quality, thereby providing insights into the early impact on male reproductive function.

ELIGIBILITY:
Inclusion Criteria:

* Male
* PCR on nasopharyngeal swab positive for SARS-CoV-2
* Age: ≥ 18y - ≤ 50y
* Signed informed consent
* When undergoing ART treatment: ICSI treatment

Exclusion Criteria:

* Negative test of SARS-CoV-2 on nasopharyngeal swab sample
* History of immunosuppression
* Impossibility to deliver a semen sample at UZ Brussel on a weekly base
* When undergoing ART treatment: IVF treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
detection of SARS-CoV-2 in the semen | within 7 days after positive testing for SARS-CoV-2
  detection of SARS-CoV-2 in the semen of men positive for SARS-CoV-2 on nasopharyngeal swab

SECONDARY OUTCOMES:
duration of SARS-CoV-2 presence in semen | from first positive semen testing until first negative semen testing, upto 15 weeks
  in case of a positive SARS-CoV-2 semen sample, for how long stays the virus present in semen
semen viscosity | from first until last semen analysis, upto 15 weeks
  viscosity of semen will be assessed macroscopically
semen volume | from first until last semen analysis, upto 15 weeks
  semen volume
semen pH | from first until last semen analysis, upto 15 weeks
  semen pH
Sperm motility | from first until last semen analysis, upto 15 weeks
  Sperm motility assesment, according to the WHO guidelines of 2010
Sperm morphology | from first until last semen analysis, upto 15 weeks
  Sperm morphology assesment, according to the WHO guidelines of 2010
Sperm density | from first until last semen analysis, upto 15 weeks
  Sperm density assesment, according to the WHO guidelines of 2010

CONTACTS AND LOCATIONS:
Overall Officials: Michael De Brucker, MD PHD, Principal Investigator — UZ Brussels
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li D, Jin M, Bao P, Zhao W, Zhang S. Clinical Characteristics and Results of Semen Tests Among Men With Coronavirus Disease 2019. JAMA Netw Open. 2020 May 1;3(5):e208292. doi: 10.1001/jamanetworkopen.2020.8292. PMID 32379329